CLINICAL TRIAL: NCT03651648
Title: Apnea Treatment in Premature Infants Using an Automatic Vibro-tactile Stimulator Triggered by the Detection of Apnea-bradycardia.
Acronym: SENSITACT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 35RC16_9894_SENSITACT
Record Dates: First submitted 2018-07-18; First posted 2018-08-29 (Actual); Last update posted 2023-11-27 (Actual); Status verified 2023-11

CONDITIONS: Apnea of Prematurity
Keywords: apnea; prematurity; kinesthetic stimulation
MeSH Terms: conditions — Apnea; Premature Birth

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SENSITACT System ON (Experimental): As soon as the early signs of an apnea-bradycardia are detected, the SENSITACT controller sends a trigger signal to the PASITHEA stimulator that immediately activates kinesthetic stimulation
  Interventions: Device: SENSITACT System
- SENSITACT System OFF (Sham Comparator): The SENSITACT controller doesnt send any trigger signal to the PASITHEA stimulator even if an early sign of an apnea-bradycardia is detected.
  Interventions: Device: SENSITACT System

INTERVENTIONS:
Device: SENSITACT System — the activated stimulation (ON period of 6 hours) will be hidden from the care team, who will continue the care according to the usual procedures (blind treatment).
  Other Names: Actived stimulation
  Arms: SENSITACT System ON
Device: SENSITACT System — the desactivated stimulation (OFF period of 6 hours) will be hidden from the care team, who will continue the care according to the usual procedures (blind treatment).
  Other Names: desactivated stimulation
  Arms: SENSITACT System OFF

SUMMARY:
The goal of the SENSITACT system is to activate an adaptive kinesthetic stimulation to treat apnea-bradycardia events on preterm infants, while minimizing deleterious effects, in particular arousals that can be due either to respiratory efforts or to kinesthetic stimulation itself. This novel system will provide an alternative treatment to apnea-bradycardia, with improved patient comfort and autonomy. In particular, it may become a complementary solution for the current treatments (Manual stimulation by caregivers, continuous or intermittent nasal positive pressure ventilation and methylxanthine therapies) that do not appear to be optimal and usually only allow a partial reduction in the number and severity of apneas.

DETAILED DESCRIPTION:
The main hypothesis behind the SENSITACT system is that kinesthetic stimulation can terminate apneas-bradycardias with minimal patient arousal. The aim is to stimulate mechanoreceptors through the skin by kinesthetic stimulation on the lower abdominal zone. This is a region of the body that is covered with Pacinian corpuscles, a very sensitive kind of mechanoreceptors, which respond to rapid vibrations on the skin (200-300 Hz). Vibro-tactile stimulation of these mechano-receptors will trigger a reaction typical of the startle reflex. This reflex causes 1) an immediate myotonic reaction and 2) a widespread autonomic response. The former should have a direct effect on obstructive respiratory disorders with an increase in chin muscle tones within 80 to 100 ms. The latter should act on central respiratory disorders, with activation of the sympathetic nervous system. Since both responses are mediated via sub-cortical nervous center, it is expected that patient arousal will be limited. Preliminary clinical studies on adult patients conducted by LTSI, Sorin CRM and CHU de Grenoble (Skin&SAS, HYPNOS, EKINOx), that have used the same PASITHEA stimulation device have confirmed activation of the sympathetic nervous system and a significant reduction in the duration of apnea or hypopnea events, while no differences were observed on patients' sleep architecture.

The SENSITACT system is able to detect apneas-bradycardias in real-time, so that kinesthetic stimulation can be triggered to stop respiratory disorders very early during the event. Detection is performed within the SENSITACT controller station that receives data from all sensors connected to the Patient Monitor in real-time. As soon as the early signs of an apnea-bradycardia are detected, the SENSITACT controller sends a trigger signal to the PASITHEA stimulator that immediately activates kinesthetic stimulation.

Kinesthetic stimulation is stopped when a normal condition (normal cardiac rhythm) is detected or when a maximum number of stimulation pulses have been reached.

ELIGIBILITY:
Inclusion Criteria:

* written informed consent,
* Premature infants,

  * born to a term less than 34 weeks of amenorrhea (AS),
  * Age less than 36 weeks post-menstrual age,
  * With a postnatal age greater than 4 days,
  * caffeine treated, for at least 36 hours,
  * Presenting episodes of bradycardia apnea significant (>10 sec with bradycardia <100 bpm or SaO2<80%) with an interval of less than 6 hours between two episodes observed in the 24 hours preceding inclusion.

Exclusion Criteria:

* Major congenital neurological abnormalities,
* Congenital abnormalities of the respiratory tracts,
* HIV grade 3 or 4,
* Periventricular leukomalacia,
* Invasive ventilation and non-invasive ventilation in NAVA mode,
* Cyanogenic malformative heart disease,
* Sepsis diagnosed in the 4 days prior to registration (CRP> 10mg / L),
* maternal addiction during pregnancy,
* Father and / or mother legally protected (under judicial protection, guardianship or supervision).

Ages: 34 Weeks to 36 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Estimated)
Dates: Start 2019-10-18 (Actual); Primary Completion 2024-01-02 (Estimated); Study Completion 2024-07-02 (Estimated)

PRIMARY OUTCOMES:
Cumulative duration of apnea-bradycardia | 12 hours (H12)
  Cumulative duration of apnea-bradycardia over a period of 6 hours with stimulation activated or not.

SECONDARY OUTCOMES:
Distribution of bradycardia durations | 12 hours (H12)
  A bradycardia is defined by an acute event lasting at least 5 seconds with a decrease in heart rate of more than 33% of the basal heart rate (median of heart measured on 5-min stationary periods during quiet sleep).
  The distribution of the durations will be quantified in terms of median, IQR and distribution curve
Depth of bradycardia | 12 hours (H12)
  A bradycardia is defined by an acute event lasting at least 5 seconds with a decrease in heart rate of more than 33% of the basal heart rate (median of heart measured on 5-min stationary periods during quiet sleep).
  The depth of bradycardia will be measured by the area under the curve with the upper limit of the curve defined by the value of "basal heart rate-33%" and expressed in beats/min*sec The distribution of the depth of bradycardias will be quantified in terms of median, IQR and distribution curve
Depth of desaturations | 12 hours (H12)
  The depth of desaturation will be measured by the area under the curve with the upper limit of the curve set at a Saturation of 80% The distribution of the depth of desaturations will be quantified in terms of median, IQR and distribution curve
Caregiver interventions | 12 hours (H12)
  The number of caregiver interventions associated with a cardio-respiatory event will be quantified and expressed in number/hour
Cardiorespiratory parameters in response to stimulation | 6 hours (H6)
  The delay between the initiation of stimulation and the first breath will be measured and expressed in median IQR The delay between the initiation of stimulation and the normalization of heart rate above the limit of "basal heart rate-33%" will be measured and expressed in median IQR The delay between the initiation of stimulation and the observation of a Saturation above 80% will be measured and expressed in median IQR
Premature's sleep-wake cycles | 12 hours (H12)
  Duration of the stages identified

CONTACTS AND LOCATIONS:
Overall Officials: Patrick PLADYS, Pr, Principal Investigator — Rennes University Hospital
Locations (1):
- CHU de Rennes, Rennes, France

IPD SHARING:
Plan to Share IPD: No